CLINICAL TRIAL: NCT03209687
Title: Human Menopausal Gonadotropin as a Novel Addition to Luteal Phase Support in Down-regulated ICSI Cycles (RCT)
Brief Title: The Value of Addition of Human Menopausal Gonadotropin Drug Following Oocytes Retrieval in IVF Cycles
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdel-Maguid Ramzy, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3778
Record Dates: First submitted 2017-07-04; First posted 2017-07-06 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Menotropins; hMG-IBSA

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Human menopausal gonadotropin (HMG) (Experimental): This group will take daily subcutaneous 75 IU (international unit) of human menopausal gonadotropin (HMG) in addition to the usual luteal phase support from the day of ovum pickup and will be continued for 2 weeks
  Interventions: Drug: human menopausal gonadotropin
- Routine care (No Intervention): This group will receive the routine care for luteal phase support

INTERVENTIONS:
Drug: human menopausal gonadotropin — Merional injections will be given to participants after ovum pickup in in-vitro fertilization cycles
  Other Names: Merional
  Arms: Human menopausal gonadotropin (HMG)

SUMMARY:
The aim of this study is to test the hypothesis that addition of daily small dose of human menopausal gonadotropin (HMG) drug following oocytes retrieval could improve the fertility outcome in women undergoing in-vitro fertilization

DETAILED DESCRIPTION:
The study will be conducted in the IVF unit of Cairo University. Females undergoing ICSI cycles in the age between 20 and 40 years will be allocated to one of 2 groups. Long agonist protocol will be used. Allocation to either one of 2 groups will be done on the day of oocytes retrieval. The first group will take (in addition to the routine care) daily human menopausal gonadotropin drug injection for 2 weeks. The second group will receive the routine care.

ELIGIBILITY:
Inclusion Criteria:

* Females undergoing Intra-Cytoplasmic Sperm Injection (ICSI) cycles
* Age between 20 and 40 years

Exclusion Criteria:

* Females who have high response (estradiol at time of ovulation trigger is > 5000 pg/ml or more than 15 oocytes are retrieved)

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2017-07-06 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | This outcome will be calculated 2 years after enrollment of the first patient in the study
  The live birth rate will be calculated by a statistician for each group

SECONDARY OUTCOMES:
Clinical pregnancy rate | This outcome will be calculated 2 years after enrollment of the first patient in the study
  The clinical pregnancy rate will be calculated by a statistician for each group
Implantation rate | This outcome will be calculated 2 years after enrollment of the first patient in the study
  The implantation rate will be calculated by a statistician for each group
Miscarriage rate | This outcome will be calculated 2 years after enrollment of the first patient in the study
  The miscarriage rate will be calculated by a statistician for each group

CONTACTS AND LOCATIONS:
Overall Officials: Abdelmaguid Ramzy, M.D., Principal Investigator — Cairo University; Eman Omran, M.D., Study Director — Cairo University
Locations (1):
- Department of Obstetrics and Gynecology, Kasr Al-Ainy hospital, Cairo, Greater Cairo, Egypt